CLINICAL TRIAL: NCT03838159
Title: A Randomized Phase II Study of Neo-adjuvant Chemo/Immunotherapy Versus Chemotherapy Alone for the Treatment of Locally Advanced and Potentially Resectable Non-small Cell Lung Cancer (NSCLC) Patients.
Brief Title: NADIM II: Neo-Adjuvant Immunotherapy
Acronym: NADIMII
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP 18/02_NADIM II; 2018-004515-45 (EudraCT Number)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Inmunotherapy; Resectable stage IIIA; Adjuvant treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Neo-Adjuvant Immunotherapy (Experimental): * Neoadjuvant treatment (200 mg/m3 Paclitaxel+ AUC5 Carboplatin+ 360 mg Nivolumab) will start within 1-3 days from randomisation. 3 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) prior to surgery. Before surgery a tumor assessment will be done. Patients must leave the study if there is evidence of progression. Patients with stable disease or partial response may be considered for surgery.
  * Surgery: Surgery must be done within the 3rd-4th week (+7 days) from day 21 cycle 3 of neoadjuvant treatment (day 42-49 after day 1 of cycle 3) .
  * Adjuvant treatment:Nivolumab: 480 mg Q4W (+/- 3 days) for 6 months (6 cycles). Patients that are R0 confirmed by surgical pathology evaluation will receive the first adjuvant administration within the 3rd to 8th week (+ 7 days) from surgery and for 6 months.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Nivolumab
- Control: Neo-Adjuvant Chemotherapy (Active Comparator): * Neoadjuvant treatment (200mg/m3 Paclitaxel+ AUC5 Carboplatin). It will start within 1-3 days from randomisation. 3 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) prior to surgery. Before surgery a tumor assessment will be done. Patients must leave the study if there is evidence of progression. Patients with stable disease or partial response may be considered for surgery.
  * Surgery: Surgery must be done within the 3rd-4th week (+7 days) from day 21 cycle 3 of neoadjuvant treatment (day 42-49 after day 1 of cycle 3)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel must be administered by infusion over 3 hours in dextrose (D5W) or normal saline (NS). The concentration must not exceed 1.2 mg/ml.
  The infusions must be mixed as soon as possible before the start of each infusion since the stability of paclitaxel beyond 24 hours is not known.
  In-line filtration is obligatory since a small number of fibers within the acceptable limits of the USP Particulate Matter Test for LVP have been reported. Cellulose acetate filters of 0.22-micron pore size (such as IVEX II) can be used. The solution that shows excessive particulate matter must be rejected.
  Other Names: Taxol
Drug: Carboplatin — Carboplatin must be administered at the end of the Paclitaxel infusion
  Other Names: Paraplatin
Drug: Nivolumab — Nivolumab is a soluble protein consisting of 4 polypeptide chains, which include 2 identical heavy chains and 2 identical light chains.
  The administration of nivolumab infusion must be completed within 24 hours of preparation.
  Other Names: Opdivo
  Arms: Experimental: Neo-Adjuvant Immunotherapy

SUMMARY:
This is an open-label, randomised, two-arm, phase II, multi-centre clinical trial.

90 patients will be enrolled in this trial to examine the pathological Complete Response defined as the absence of residual tumor in lung and lymph nodes comparing patients treated with chemo-immunotherapy versus chemotherapy alone.

DETAILED DESCRIPTION:
This is an open-label, randomised, two-arm, phase II, multi-centre clinical trial.

Patients randomised to the experimental arm will receive Nivolumab 360mg + Paclitaxel 200mg/m2 + Carboplatin AUC5 for 3 cycles every 21 days as neoadjuvant treatment followed by surgery and 6 months of adjuvant treatment with Nivolumab 480 mg Q4W. Patients randomized to the control arm will receive Paclitaxel 200mg/m2 + Carboplatin AUC5 for 3 cycles every 21 days followed by surgery.

The primary objective is pathological Complete Response (pCR) defined as the absence of residual tumor in lung and lymph nodes comparing patients treated with chemo-immunotherapy versus chemotherapy alone.

Patient accrual is expected to be completed within 3 years excluding a run-in-period of 3 months. Treatment and follow-up are expected to extend the study duration to a total of 8.5 years. Patients will be followed 5 years after adjuvant treatment or surgery. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated patients with histologically- or cytologically- documented NSCLC who present stage IIIA disease (according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) and also, potentially resectable locally advanced NSCLC patients' stage IIIB with T3N2 disease according to 8th edition can be included.

   * PET/CT including IV contrast (CT of diagnostic quality) will be performed at baseline (28 days +10 before randomization)
2. Tumor should be considered resectable before study entry by a multidisciplinary team
3. ECOG (Performance status) 0-1
4. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization.

   i. Neutrophils ≥ 1500×109/L ii. Platelets ≥ 100 x×109/L iii. Hemoglobin > 9.0 g/dL iv. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min v. AST/ALT ≤ 3 x ULN vi. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) vii. The patients need to have a forced expiratory volume (FEV1) ≥ 1.2 liters or >40% predicted value viii. INR/APTT within normal limits
5. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention
6. Patients aged > 18 years
7. Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before randomization.
8. All sexually active men and women of childbearing potential must use an effective contraceptive method (two barrier methods or a barrier method plus a hormonal method) during the study treatment and for a period of at least 12 months following the last administration of trial drugs
9. Patient capable of proper therapeutic compliance and accessible for correct follow-up
10. Measurable or evaluable disease (according to RECIST 1.1 criteria)

Exclusion Criteria:

1. All patients carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene.
2. Patients with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement or unexpected conditions of recurrence in the absence of an external trigger are allowed to be included.
3. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
4. Patients with a history of interstitial lung disease cannot be included if they have symptomatic ILD (Grade 3-4) and/or poor lung function. In case of doubt please contact trial team.
5. Patients with other active malignancy requiring concurrent intervention and/or concurrent treatment with other investigational drugs or anti-cancer therapy
6. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
7. Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information
8. Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
9. Patients with positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
10. Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
11. Patients with history of allergy to study drug components excipients
12. Women who are pregnant or in the period of breastfeeding
13. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the pathological complete response (pCR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 45 months.
  The pathological complete response is defined as the absence of residual tumor in lung and lymph nodes in patients treated with chemo-immunotherapy versus patients treated with chemotherapy alone.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Hospital Puerta del Hierro
Locations (25):
- Spain (25):
  - ICO Badalona, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital General de Alicante, Alicante
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario de Málaga, Málaga
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Provencio M, Nadal E, Gonzalez-Larriba JL, Martinez-Marti A, Bernabe R, Bosch-Barrera J, Casal-Rubio J, Calvo V, Insa A, Ponce S, Reguart N, de Castro J, Mosquera J, Cobo M, Aguilar A, Lopez Vivanco G, Camps C, Lopez-Castro R, Moran T, Barneto I, Rodriguez-Abreu D, Serna-Blasco R, Benitez R, Aguado de la Rosa C, Palmero R, Hernando-Trancho F, Martin-Lopez J, Cruz-Bermudez A, Massuti B, Romero A. Perioperative Nivolumab and Chemotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Aug 10;389(6):504-513. doi: 10.1056/NEJMoa2215530. Epub 2023 Jun 28. PMID 37379158
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org